CLINICAL TRIAL: NCT02459431
Title: Impact of Needle Size on the Diagnosis of Sarcoidosis by Endobronchial Ultrasound Guided Transbronchial Needle Aspiration: Randomized Trial Comparing 21-Gauge and 22-Gauge Needles
Brief Title: RCT Comparing 21 and 22 G Needle in the Diagnosis of Sarcoidosis by EBUS TBNA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Ritesh Agarwal, Additional professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: PGIMERpulmoIndia
Record Dates: First submitted 2015-05-26; First posted 2015-06-02 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2017-01

CONDITIONS: Sarcoidosis
MeSH Terms: conditions — Sarcoidosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 21G needle group (Active Comparator): 21 gauge endobronchial ultrasound guided transbronchial aspiration needle ( Vizishot, Olympus ) would be used to perform endobronchial ultrasound guided Transbronchial needle aspiration
  Interventions: Other: 21 G needle group
- 22G needle group (Active Comparator): 22 gauge endobronchial ultrasound guided transbronchial aspiration needle ( Vizishot, Olympus ) would be used to perform endobronchial ultrasound guided Transbronchial needle aspiration
  Interventions: Other: 22 G needle group

INTERVENTIONS:
Other: 21 G needle group — Patients with a clinico radiologic suspicion of sarcoidosis will undergo endobronchial ultrasound guided transbronchial needle aspiration with 21 G needle, by random assignment
  Arms: 21G needle group
Other: 22 G needle group — Patients with a clinico radiologic suspicion of sarcoidosis will undergo endobronchial ultrasound guided transbronchial needle aspiration with 22 G needle, by random assignment
  Arms: 22G needle group

SUMMARY:
Randomized controlled trial to determine the efficacy of different needles sizes (22G and 21G) used in endobronchial ultrasound guided transbronchial needle aspiration

DETAILED DESCRIPTION:
Among the bronchoscopic techniques in diagnosis of sarcoidosis, transbronchial needle aspiration (TBNA) of lymph nodes has emerged as a particularly useful supplement to the previously known endobronchial and transbronchial biopsies. The efficacy and safety of conventional TBNA is well established. With improvements in technology, the last decade has seen the use of convex probe endobronchial ultrasonography (EBUS) to guide TBNA under direct vision. This technique is a minimally invasive alternative to mediastinoscopy, further it offers additional advantage of choosing the appropriate node for sampling on the basis of their echogenicity. Studies subsequently have demonstrated the superiority of EBUS TBNA over conventional TBNA.

Once the role of TBNA in diagnostic bronchoscopy was established, technical aspects of the procedure became the topic of research. Needle size used in TBNA is one such important factor. Apparently, larger the needle, better the tissue yield and hence improved diagnostic capability. Conventional TBNA is usually performed with a 19G needle, though varying sizes have been used in different studies (18, 21, 22, 26G). On the other hand, EBUS-TBNA is performed with a 22G needle. More recently 21G needles are being used for the same purpose. There have been conflicting reports in literature, when these two needle sizes have been compared with regards to the adequacy of the sample, accuracy of diagnosis and the rate of complications. Moreover, the above studies undertaken so far were done from centers where malignancy was the predominant diagnosis. Whether the needle size used during EBUS TBNA has any impact on diagnosing benign diseases like sarcoidosis is still not clear, hence this study was planned. The investigators hypothesize that performing EBUS-TBNA using 21G needles may enable identification of intact compact granulomas in sarcoidosis, and hence a better diagnostic yield than using a 22G needle.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Clinicoradiological suspicion of sarcoidosis where endobronchial ultrasound guided transbronchial needle aspiration is contemplated
* Enlarged hilar and mediastinal lymph nodes >10 mm (any axis) on computed tomography of the chest

Exclusion Criteria:

* Hypoxemia (SpO2 <92%) on inspired fraction of oxygen 0.3
* Treatment with systemic glucocorticoids for more than 2 weeks in the preceding three months
* Diagnosis of sarcoidosis possible with another minimally invasive technique such as skin biopsy or peripheral lymph node biopsy
* Failure to provide informed consent

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2013-12; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
The diagnostic yield of EBUS TBNA with 21G and 22G needle in patients with a final diagnosis of sarcoidosis will be assessed for any difference between the two | outcome assessed 6 months following enrollment of the last patient

SECONDARY OUTCOMES:
Adequacy of samples | 0, 7, 180 days of inclusion
  Samples will be considered adequate if the cytologic assessment shows lymphocytes and or definite if the specimen shows epithelioid cell granulomas or collection of epithelioid cells with a giant cell (or asteroid body or Schaumann body). The samples will be classified as: diagnostic, adequate but non-diagnostic, non-diagnostic and not adequate, no specimen
Complications | 0, 7 , 180 days of inclusion
  Complications encountered with both needle sizes will be compared if there is any difference in the rate of complications

CONTACTS AND LOCATIONS:
Overall Officials: Ritesh Agarwal, DM, Principal Investigator — Additional professor
Locations (1):
- Postgraduate Institute of Medical Education and Research, Chandigarh, Chandigarh, India